CLINICAL TRIAL: NCT02884999
Title: Management of Bleeding and Coagulopathy in Trauma and Compliance to European Trauma Guidelines
Acronym: APP
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: APP
Record Dates: First submitted 2016-08-19; First posted 2016-08-31 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Wounds and Injury; Bleeding
Keywords: trauma; bleeding; coagulopathy; guidelines compliance; recommendation; transfusion
MeSH Terms: conditions — Wounds and Injuries; Hemorrhage; Hemostatic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- severe trauma patients: Severe trauma patients admitted to the site in the first 24 hours

SUMMARY:
This cohort study describes the epidemiology of trauma patients and their management in a French academic trauma center. It also aims to determine what recommendations from the European trauma guidelines is applied in routine.

DETAILED DESCRIPTION:
Severe trauma is responsible for more than 5 millions of deaths annually worldwide. Haemorrhagic shock secondary to uncontrolled bleeding is the leading cause of preventable death in this population, making bleeding and coagulopathy treatment a key element of the early phase of trauma management. European trauma guidelines have been developed to help clinicians in severe trauma management and improve bleeding and coagulopathy treatment in this population. Investigating who these guidelines are followed in routine is crucial to identify opportunities to improve early management of bleeding severe trauma patients.

ELIGIBILITY:
Inclusion Criteria:

* Trauma patients with injury severity score equal to or higher than 16 year old admitted to the Brest academic trauma centre within the 24 hours following the trauma

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Severe trauma patients
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2015-05; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Number of patients treated as per studied guidelines | first 24 hours of trauma management

CONTACTS AND LOCATIONS:
Overall Officials: Cécile Aubron, Study Director — CHRU de Brest
Locations (1):
- CHRU de BRest, Brest, France

IPD SHARING:
Plan to Share IPD: No